CLINICAL TRIAL: NCT03432598
Title: A Phase II, Open-Label, Multi-Cohort Study to Investigate the Preliminary Antitumor Activity, Safety, and Pharmacokinetics of the Anti-PD-1 Monoclonal Antibody BGB-A317 in Combination With Chemotherapy as First-Line Treatment in Chinese Subjects With Locally Advanced or Metastatic Lung Cancer
Brief Title: Anti-PD-1 in Combination With Chemotherapy as First-Line Treatment to Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-206; CTR20170361 (Registry Identifier: Center for drug evaluation, CFDA)
Record Dates: First submitted 2018-02-08; First posted 2018-02-14 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Locally Advanced Lung Cancer; Metastatic Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — tislelizumab; Paclitaxel; Gemcitabine; Etoposide; Pemetrexed; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Non-squamous NSCLC (Experimental): Day 1 of each 21-day (3 weeks) cycle: Tislelizumab + pemetrexed + cisplatin 75 mg/m²/day IV (or carboplatin AUC 5).
  Pemetrexed plus cisplatin (or carboplatin) should be given for up to 4 cycles.
  Following either completion of or discontinuation from chemotherapy, tislelizumab will be continued as scheduled, if clinically appropriate. Pemetrexed maintenance after completion of doublet chemotherapy is permitted.
  Interventions: Drug: Tislelizumab; Drug: Pemetrexed; Drug: Cisplatin; Drug: Carboplatin
- Squamous NSCLC Cohort A (Experimental): Tislelizumab every 3 weeks (Q3W) + paclitaxel + cisplatin (or carboplatin), Q3W.
  Paclitaxel plus cisplatin (or carboplatin) will be administered for 4-6 cycles.
  Following either completion of or discontinuation from chemotherapy, tislelizumab will be continued as scheduled, if clinically appropriate.
  Interventions: Drug: Tislelizumab; Drug: Paclitaxel; Drug: Cisplatin; Drug: Carboplatin
- Squamous NSCLC Cohort B (Experimental): Tislelizumab Q3W on Day 1 + gemcitabine on Day 1 and Day 8 + cisplatin IV (or carboplatin) on Day 1.
  Gemcitabine plus cisplatin (or carboplatin) will be administered for 4-6 cycles.
  Following either completion of or discontinuation from chemotherapy, tislelizumab will be continued as scheduled, if clinically appropriate.
  Interventions: Drug: Tislelizumab; Drug: Gemcitabine; Drug: Cisplatin; Drug: Carboplatin
- SCLC (Experimental): Tislelizumab Q3W on Day 1, etoposide on Days 1, 2, and 3 + cisplatin (or carboplatin) on Day 1.
  Etoposide and cisplatin (or carboplatin) will be administered for 4-6 cycles.
  Following either completion of or discontinuation from chemotherapy, tislelizumab will be continued as scheduled, if clinically appropriate.
  Interventions: Drug: Etoposide; Drug: Cisplatin; Drug: Carboplatin

INTERVENTIONS:
Drug: Tislelizumab — Administered 200 mg intravenously (IV) as specified in the treatment arm
  Other Names: BGB-A317
  Arms: Non-squamous NSCLC; Squamous NSCLC Cohort A; Squamous NSCLC Cohort B
Drug: Paclitaxel — Administered 175 mg/m² IV as specified in the treatment arm
  Arms: Squamous NSCLC Cohort A
Drug: Gemcitabine — Administered 1250 mg/m² IV as specified in the treatment arm
  Arms: Squamous NSCLC Cohort B
Drug: Etoposide — Administered 100 mg/m2 IV as specified in the treatment arm
  Arms: SCLC
Drug: Pemetrexed — Administered 500 mg/m² IV as specified in the treatment arm
  Arms: Non-squamous NSCLC
Drug: Cisplatin — Administered 75 mg/m²/day IV as specified in the treatment arm
Drug: Carboplatin — Administered AUC 5 as specified in the treatment arm

SUMMARY:
This is a Phase II, open-label, 4-cohort study of the monoclonal antibody BGB-A317 in combination with standard platinum-based chemotherapy in participants with advanced NSCLC or SCLC. The 4 cohorts will be enrolled concurrently including non-squamous NSCLC Cohort, squamous NSCLC Cohort A, squamous NSCLC Cohort B and SCLC Cohort. Participants with a mixed adenocarcinoma and squamous cell NSCLC will be allocated to one of the NSCLC cohorts based on the predominant histopathological profile. (e.g., participants with adenocarcinoma component accounting for > 50% will be allocated to non-squamous NSCLC cohort.). Participants with squamous NSCLC will be sequentially enrolled into either of the 2 squamous NSCLC cohorts by the trial stage i.e. the sequence of the enrollment for the squamous NSCLC cohorts will be as Cohort A safety run-in Stage, followed by Cohort B safety run-in Stage, Cohort A dose-expansion stage and Cohort B dose-expansion Stage.

ELIGIBILITY:
Key Inclusion Criteria:

1. Male or female, aged 18-75 years on the day of signing informed consent.
2. Have histologically or cytologically confirmed locally advanced or metastatic non-squamous NSCLC, squamous NSCLC, or extensive-stage SCLC.

   Note: Participants with mixed adenosquamous carcinoma may also be enrolled on a case-by-case basis after discussion with the medical monitors.
3. Have had no prior systemic therapy for advanced or metastatic disease. Prior neoadjuvant/adjuvant therapy or chemoradiation therapy with curative intent should have been completed at least 6 months prior to documentation of recurrence of disease.
4. Participants must be able to provide fresh or archival tumor tissues (formalin-fixed paraffin-embedded [FFPE] blocks or at least 10 unstained FFPE slides) with an associated pathological report.

Key Exclusion Criteria:

1. Participants with a sensitizing mutation in EGFR gene or an ALK fusion oncogene (specifically for participants with non- squamous NSCLC). Participants with unknown mutation/fusion status of EGFR and/or ALK must take the respective test at the investigational sites (or other designated sites) prior to enrolment.
2. Prior malignancy active within the previous 2 years exceptions include the tumor under investigation in this trial, and locally recurring cancers that have undergone curative treatment, such as resected basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix or breast
3. Prior therapies targeting PD-1, PD-L1 or PD-L2

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2017-08-24 (Actual); Primary Completion 2019-02-25 (Actual); Study Completion 2020-12-21 (Actual)

PRIMARY OUTCOMES:
The objective response rate (ORR) as assessed by the Investigator according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 | Up to 4 years

SECONDARY OUTCOMES:
The incidence and severity of adverse events (AEs) according to NCI-CTCAE Version 4.03 | Up to 4 years
Duration of Response (DoR) - defined as the time from the first determination of a confirmed objective response according to RECIST v1.1 until the first documentation of progression or death, whichever comes first | Up to 4 years
Progression-Free Survival (PFS) - defined as the time from the date of first dose of study treatment to the date of first documentation of disease progression using RECIST v1.1 or death, whichever occurs first | Up to 4 years
Disease Control Rate (DCR) - defined as the proportion of participants who achieve CR, PR and SD using RECIST v1.1 | Up to 4 years
Pharmacokinetic evaluations of BGB-A317 in combination with chemotherapy: including but not limited to Ctrough | Up to 4 years
Anti-BGB-A317 antibody: immunogenic responses to BGB-A317 will be assessed to determine occurrence of anti-drug antibody. | Up to 4 years
The abnormality of laboratory tests according to NCI CTCAE Version 4.03 | Up to 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Jie Wang, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Locations (7):
- China (7):
  - Cancer Hospital Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Beijing Chest Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - Jilin Cancer Hospital, Changchun, Jilin
  - The First Hospital of Jilin University, Changchun, Jilin

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Wang Z, Zhao J, Ma Z, Cui J, Shu Y, Liu Z, Cheng Y, Leaw SJ, Wu Y, Ma Y, Tan W, Ma X, Zhang Y, Wang J. A Phase 2 Study of Tislelizumab in Combination With Platinum-Based Chemotherapy as First-line Treatment for Advanced Lung Cancer in Chinese Patients. Lung Cancer. 2020 Sep;147:259-268. doi: 10.1016/j.lungcan.2020.06.007. Epub 2020 Jun 20. PMID 32769013